CLINICAL TRIAL: NCT05086354
Title: Examining a Fast Movement Approach to Pediatric Therapy Intervention in Children and Adolescents That Have Completed Medical Treatment for Acute Lymphoblastic Leukemia
Brief Title: Examining a Training Program for for Acute Lymphoblastic Leukemia Childhood Cancer Survivors
Acronym: JUMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, victoria marchese, Associate Professor, Chair, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00078339
Record Dates: First submitted 2021-09-27; First posted 2021-10-20 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Childhood Cancer
Keywords: physical therapy; functional mobility
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Feasibility study
Masking Description: the physical therapist performing the baseline and post-training does not have involvement with the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One group that all receive the intervention of jumping rope. (Experimental): All participants will be in one group. Every participant receives the same intervention.
  Interventions: Behavioral: JUMP

INTERVENTIONS:
Behavioral: JUMP — Warm-up, stretching, jumping rope, cool-down

SUMMARY:
Acute lymphoblastic leukemia (ALL) is the most common pediatric malignancy, with the peak incidences occurring in children two to five years of age. Children with ALL received neurotoxic chemotherapy agents for two to three years that causes decreased distal muscle strength and poor timing of muscle activation. After completion of medical treatment, ALL childhood cancer survivors (ALL CCS) are more likely to have an inactive lifestyle, resulting in life-long gross motor proficiency differences compared to their peers. ALL CCS typically do not utilize physical therapists' expertise after medical treatment has been completed. There are limited physical therapy (PT) intervention studies for ALL CCS.

DETAILED DESCRIPTION:
We are performing a feasibility study to examine a movement based intervention that utilizes fast movements through jumping rope to improve balance, coordination, movement speed, and movement agility. The abilities to generate fast movements are required to perform functional activities and for playing sports. Participants will receive five in-person PT sessions and a home program for six weeks. The goal of this research is to determine the feasibility, acceptability, and promise of a PT program that emphasizes fast movements in ALL CCS.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-17 years old
* Completed medical treatment for ALL within the past five years (1 to 60 months)
* Speak English.

Exclusion Criteria:

* Diagnosis of a neurological disorder such as cerebral palsy, Down syndrome
* Currently receiving PT services.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Gross Motor Proficiency | 20 minutes
  Bruininks-Oseretsky Test of Motor Proficiency 2nd edition (BOT-2) (subtest 4, 5, 6, 8: bilateral coordination, balance, running speed and agility, and strength). The BOT-2 is a reliable and valid norm-referenced instrument designed for children and adolescents 4-21 years old.

SECONDARY OUTCOMES:
Children's Assessment of Participation and Enjoyment (CAPE) questionnaire. | 10 minutes
  The CAPE are designed for use with children ages 6-21 years old.
electromyography (EMG) | 5 minutes
  The EMG onset will be defined by the time when the EMG burst is 3 standard deviations above the baseline muscle activity. The slope of the muscle activity, which is the linear regression line of best fit for the values between the onset of the EMG, and the peak of the EMG burst amplitude will be calculated and normalized by dividing the slope by the peak amplitude. The EMG burst slope reflects the recruitment and firing rate of motor units at the onset of the contraction, which is important for producing fast responses.
Preferences for Physical Activity for Children (PAC) | 10 minutes
  This is a survey to explore physical activity preferences of children.
Vertical Jump Height | 5 minutes
  Participants will perform five vertical jumps starting in the upright standing position with their feet on two adjacent force platforms. The instructions will be to "jump straight up as high as you can".
Peak vertical ground reaction | 5 minutes
  participant is asked to jump on the force platform. Takeoff is defined as the highest vertical ground reaction force value attained from the force time record for the takeoff phase of each jump, minus body mass
Motion Capture Analysis | 5 minutes
  The 3D motion analysis will be captured with a VICON T10 Camera with Nexus Software VICON markers will be placed on each shoe in the position of the great toe, ankle (lateral malleoli), lateral knee (proximal to the apex of the fibular head), greater trochanter of the hip, shoulder (greater tubercle of the humerus), lateral elbow (distal to lateral epicondyle), the wrist (styloid process), and head (wearing a headband).

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Marchese, PT, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine Dept. of Physical Therapy & Rehabilitation Science, Baltimore, Maryland, United States